CLINICAL TRIAL: NCT03559621
Title: Mobile-based Lifestyle Intervention in Women With Glucose Intolerance After Gestational Diabetes
Acronym: MELINDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: the Melinda study
Record Dates: First submitted 2018-05-23; First posted 2018-06-18 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Gestational Diabetes; Type 2 Diabetes Mellitus; Glucose Intolerance; Healthy Lifestyle
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: RCT with a mobile based lifestyle intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Women in the control group will receive follow-up as in normal routine with referral to primary care. They will receive an OGTT after 1 year as part of the trial.
- intervention group (Other): A mobile-based lifestyle intervention
  Interventions: Behavioral: mobile-based lifestyle intervention

INTERVENTIONS:
Behavioral: mobile-based lifestyle intervention — one face-to-face coaching within 2 weeks after randomization, monthly telephonic coaching -and continuous use of the app as needed
  Arms: intervention group

SUMMARY:
Although lifestyle modification programs have been shown to be effective in preventing diabetes in older populations, interventions in women with recent gestational diabetes (GDM) clearly need to be adapted to address their unique barriers to behavior change in order to optimize adherence. The low participating rates in many studies using individual or group sessions, reflect how difficult it is to engage women in the first years postpartum. Since women with glucose intolerance (prediabetes) have the highest risk to develop type 2 diabetes (T2DM), we designed the MELINDA pilot study, a randomized controlled trial with 1 year of follow-up to evaluate the efficacy and feasibility of a telephone -and mobile (app) based lifestyle coaching intervention in women with glucose intolerance after a recent history of GDM to promote a healthy lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or older
* GDM based on the 2013 WHO criteria
* glucose intolerance (prediabetes based on the ADA criteria) based on the 75g OGTT 6-16 weeks after delivery

Exclusion Criteria:

* diabetes;
* current use of metformin;
* normal glucose tolerance (ADA criteria);
* health limitations or treatments which would restrict the participation in the intervention trial.
* Has no smartphone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-04-14 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
weight-loss goal | 1 year
  reaching the weight-loss goal ≥5% of body weight when overweight or obese or returning to pre-gravid weight if normal BMI

SECONDARY OUTCOMES:
diabetes | 1 year
  development of type 2 diabetes based on the ADA criteria
prediabetes | 6-16 weeks postpartum
  prevalence of prediabetes based on the ADA criteria
prediabetes | 1 year postpartum
  prevalence of prediabetes based on the ADA criteria
metabolic syndrome | 1 year
  development of a metabolic syndrome based on the WHO criteria
metabolic syndrome | 6-16 weeks postpartum
  development of a metabolic syndrome based on the WHO criteria
insulin resistance Matsuda | 1 year
  insulin resistance measured by Matsuda index
insulin resistance HOMA-IR | 1 year
  insulin resistance measured by HOMA-IR
beta-cell function ISSI-2 index | 1 year
  beta-cell function measured by ISSI-2 index
beta-cell function insulinogenic index | 1 year
  beta-cell function measured by insulinogenic index
beta-cell function HOMA-B | 1 year
  beta-cell function measured by HOMA-B
weight loss | 1 year
  mean weight loss
duration breastfeeding | 1 year
  self-designed questionnaire to evaluate duration of breastfeeding
rate exclusive breastfeeding | 1 year
  self-designed questionnaire to evaluate rate of exclusive breastfeeding
quality of life | 1 year
  SF-36 questionnaire
depression | 1 year
  CES-D questionnaire
anxiety | 1 year
  STAI-6 questionnaire
motivation for behavior change | 1 year
  the TSRQ
dietary quality | 1 year
  Flemish FFQ
physical activity IPAQ | 1 year
  IPAQ questionnaire
physical activity pedometer | 1 year
  pedometer
diabetes risk perception | 1 year
  diabetes risk perception questionnaire
Sence of Coherence | 1 year
  Sence of Coherence (SOC) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Benhalima, MD PhD, Principal Investigator — UZ Leuven
Locations (7):
- Belgium (7):
  - OLV Aalst-Asse, Aalst, Oost-Vlaanderen
  - GZA, Antwerp
  - UZA, Antwerp
  - Imelda Bonheiden, Bonheiden
  - AZ Klina, Brasschaat
  - AZ Groeninge Kortrijk, Kortrijk
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Minschart C, Myngheer N, Maes T, De Block C, Van Pottelbergh I, Abrams P, Vinck W, Leuridan L, Driessens S, Mathieu C, Billen J, Matthys C, Laenen A, Bogaerts A, Benhalima K. Effectiveness of a blended mobile-based lifestyle intervention in women with glucose intolerance after a recent history of gestational diabetes (MELINDA): a 1-year, prospective, multicentre, randomised controlled trial. EClinicalMedicine. 2024 Mar 8;70:102523. doi: 10.1016/j.eclinm.2024.102523. eCollection 2024 Apr. PMID 38495521